CLINICAL TRIAL: NCT02292862
Title: Search for Maternal Microchimerism in Swollen Portal Lymph Nodes of Infants With Biliary Atresia.
Brief Title: Maternal Microchimerism in Lymph Nodes of Infants With Biliary Atresia at Time of Kasai's Operation
Acronym: K-LNMC
Status: Completed | Type: Observational
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Collaborators: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Carsten Engelmann, Head of Department, Medizinische Hochschule Brandenburg Theodor Fontane
Other Study IDs: Trial 1650 12
Record Dates: First submitted 2014-11-13; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lymph nodes from children Whole Blood from mother and infant
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MG Main Group: lymph node and blood sampling
  Interventions: Procedure: Lymph node and blood sampling

INTERVENTIONS:
Procedure: Lymph node and blood sampling — By bipolar dissection 1 portal and 1 mesenteric lymph node are removed from the infant.
  Blood (1ml) is taken from mother and infant.

SUMMARY:
Maternal microchimerism has been discussed as an etiological mechanism in infantile (perinatal) biliary atresia (BA). In Kasai's operation (resection of the liver hilum plaque followed by hepato-portoenterostomy) surgeons frequently encounter swollen portal and mesenteric lymph nodes.

Lymph nodes were sampled during Kasai' s operation and examined for maternal DNA.

DETAILED DESCRIPTION:
Upon operation of infants with non-syndromatic biliary atresia (BA, commonest form), surgeons almost invariably note the prominent finding of multiple swollen lymph nodes of up to 2 cm in size in the porta hepatis and the small bowel mesentery where they may constitute grape like complexes. Same-age infants laparotomized for other pathology commonly do not present such nodes.

Biliary atresia is a disease of the newborn which is fatal when left untreated. Histologically it corresponds to a degeneration of intra- und extra hepatic bile ducts within a in part specific inflammatory infiltrate and progressive cirrhosis.

The etiology of this rare but constant disease (1:8-1:15.000) is unknown. Currently in BA etiology research two main avenues are pursued:

1. Virally induced perinatal (auto)immune processes are suspected. An experimental form of BA can be provoked by infecting murine mothers with dsRNA-viruses e.g. Rhesus-rotaviruses or Reo-viruses while in mice, vaccination of mothers has prevented experimental BA . The importance of the γ/δ-T-cell and IL17/IL 23 pathway , for BA is currently probed. However, in groups of syngenic animals treated by the same batch of viruses BA tends to be inconstant and it is limited to extrahepatic bile ducts such as about the validity of the animal model is an issue.
2. The other direction of research does not primarily rely on experiments involving newborn animals: There are indications that during pregnancy the placental barrier may become permeable for maternal lymphocytes (e.g. by a faulty silencing of T-cell attracting chemokines in decidual stroma cells) and already in 2008 maternal lymphocytes have been demonstrated in livers of BA infants . Subsequently the phenomenon of materno-fetal microchimerism has come into focus of BA ethiology research: in the context of mixed materno-fetal immune reactions cells of maternal origin could misdirect the immature immune system of the infant into auto-immunity or act directly as effectors in a graft vs. host like fashion.

The importance of mesenteric and portal lymph nodes for maturation of the immune system during pregnancy has been reported recently . Moreover it has been demonstrated that flow the between liver and portal lymph nodes is bidirectional . In In mice the frequence of CD4+ and FoxP3+ regulatory T-cells was found to be linked to the mothers immune status. We thus hypothesized that the prominently swollen lymph nodes of BA infants which surgeons constantly encounter during Kasai's operation may hold a key to the better understanding of pathophysiological important lymphocyte trafficking mechanisms.

In the standard operation, the Kasai-operation which in a race with increasing liver cirrhosis makes sense up to an age of 4 months, the degraded rests of the major bile ducts in the liver hilus (the so called "hilar plate") are resected, A Roux y-loop is sutured onto the resection site. It shall drain any contingent bile flow from remaining bile ducts. The long term success rate of this tentative of surgical cure which is of moderate technical complexity and invasiveness is estimated to ca. 15-20%. In the remaining a partly sucess may postpone the necessity of liver transplantation. We examined in seven consecutive patients with histologically proven biliary atresia whether in periportal lymph nodes there was evidence for maternal gentic material.

Methods :

7 consecutive patients with the preoperative diagnosis of BA were included in the study. Other causes of icterus prolongatus (α1 anti-trypsin deficiency, Alagilles syndrom, PFIC etc.) had been excluded amongst the methods technical successful ERCP (5/7 patients) which showed absence of intrahepatic bile ducts.

After obtaining the parent's informed consent 2 ml EDTA whole blood were collected from mother and infant. During Kasai's operation one portal and one mesenterial lymphnode were sampled (Hannover Medical School ethical committee vote No.1650/11.12.2012. After bipolar dissection the mesenteric gaps were closed with 4-0 Vicryl sutures.

Lymph nodes were disrupted mechanically and DNA was extracted enzymatically (QIAmp Kit, Qiagen, Hilden/Germany) as described previously and normalized to 30 ug/ml.

Short tandem repeat analysis was realized with multiplex PCR for markers LIPOL, VWA, TH01, D19S253, CSF, PLA2A. FGA, D21S11, D18S51 as described. Briefly, fragment length analysis was performed an Abi Prism 310 System with GeneScan 3.11. software for comparison of mother's and infant's blood with lymph node DNA.

Genetic single nucleotide polymorphisms (SNPs) were traced by quantitative real time PCR chimerism analyses. Reactions were executed on an iCycler iQ5 real-time PCR platform (Bio-Rad) using the ABsolute QPCR Rox Mix (Thermo scientific). Custom designed primers and probes were provided by Sigma-Aldrich. Control reactions and normalization of sample DNA were performed by amplifying the albumin gene.

ELIGIBILITY:
Inclusion Criteria:

* Non-Syndromatic Form of Biliary Atresia

Exclusion Criteria:

* Syndromatic Form of Biliary Atresia
* Other Congenital Liver Disease (Like Alagilles' Syndrome)
* No liver fibrosis/cirrhosis in Histology of LIver Specimen from Routine Histology

Ages: 4 Weeks to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with newly and preoperatively diagnosed infantile Biliary Atresia of the non-syndromatic form
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Maternal DNA in offspring | 3 months
  The presence of maternal DNA in the childs blood and lymph nodes is the endpoint

SECONDARY OUTCOMES:
Serum Bilirubin | perioperatively
Composition of lymphocyte population in mesenteric lymph nodes | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Carsten R Engelmann, MD, OhD, Principal Investigator — Klinikum Brandenburg
Locations (1):
- Pediatric Surgery Department, Hanover, Lower Saxony, Germany

REFERENCES:
- [Background] Leveque L, Hodgson S, Peyton S, Koyama M, MacDonald KP, Khosrotehrani K. Selective organ specific inflammation in offspring harbouring microchimerism from strongly alloreactive mothers. J Autoimmun. 2014 May;50:51-8. doi: 10.1016/j.jaut.2013.10.005. Epub 2013 Nov 20. PMID 24268809
- [Background] Willasch A, Schneider G, Reincke BS, Shayegi N, Kreyenberg H, Kuci S, Weber G, Van Der Reijden B, Niethammer D, Klingebiel T, Bader P. Sequence polymorphism systems for quantitative real-time polymerase chain reaction to characterize hematopoietic chimerism-high informativity and sensitivity as well as excellent reproducibility and precision of measurement. Lab Hematol. 2007;13(3):73-84. PMID 17984038
- [Derived] Engelmann C, Maelzer M, Kreyenberg H. Absence of Maternal Microchimerism in Regional Lymph Nodes of Children With Biliary Atresia. J Pediatr Gastroenterol Nutr. 2016 Jun;62(6):804-7. doi: 10.1097/MPG.0000000000001093. PMID 26756872